CLINICAL TRIAL: NCT06227702
Title: Vexus-guided Fluid Management in Patients With Septic Shock After the Resuscitation Phase
Acronym: VEXUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: BRICNET - Brazilian Research in Intensive Care Network (Unknown)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEXUS
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Critically Ill Patients; Septic Shock
Keywords: vexus; fluid management; deresuscitation; deaccumulation
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VeXus (Active Comparator): Patients in the intervention arm wil be assessed by VeXus. Patients without signs of venous congestion (VeXus = 0) will be observed every 6 hours. In patients with VeXus ≥1, continuous infusion of intravenous furosemide will be initiated. During the first 48 hours, furosemide infusion will be adjusted according to VeXus . All other aspects of care will be managed according to routine unit protocols
  Interventions: Other: Fluid management according to Venous Excess Ultrasound (VExUS) Score
- Usual care (No Intervention): The usual care arm will follow the management protocols of the unit which are based in the Surviving Sepsis Campaign guidelines.

INTERVENTIONS:
Other: Fluid management according to Venous Excess Ultrasound (VExUS) Score — Management of furosemide intravenous infusion according to VeXus results
  Arms: VeXus

SUMMARY:
It is well recognized the association between fluid volume administered and positive fluid balance with adverse outcomes . Active fluid removal is widely practiced in an attempt to mitigate this potential damage. However, it is not clear which is the best approach for the post-resuscitation phase in critically ill patients. In this context, Point-of-Care ultrasound (POCUS) through Venous Excess Ultrasound (VExUS) would allow the assessment of the degree of venous congestion, through the visualization of vascular anatomy and blood velocity using Doppler, being potentially useful to guide fluid removal. The investigators will evaluate whether fluid management after the initial phase of VExUS-guided resuscitation is able to improve outcomes compared to usual therapy in patients with septic shock.

This is a single center, prospective, open and randomized clinical study in which patients admitted to intensive care will be included after the first 24 hours of resuscitation. A total of 200 patients will be randomized either to volume management guided by VExUS or to the standard therapy arm as per usual practice.

DETAILED DESCRIPTION:
All patients hospitalized or admitted to the intensive care unit with septic shock will be screened for eligibility. Patients will be randomized using an electronic system (RedCap) to receive or not the intervention.

After 24 hours of shock onset, patients without hypoperfusion after informed consent will be allocated into two groups. In intervention arm wil be assessed by VeXus. Patients without signs of venous congestion (VeXus = 0) will continue to be observed every 6 hours. In patients with VeXus ≥1, continuous infusion of intravenous furosemide will be initiated. During the first 48 hours after inclusion in the study, patients will be evaluated for the intervention every 6 to 8 hours: Time 1 (T1) at randomization, T2 after 6 hours of T1, T3 after 6 hours of T2 and every 6 to 8 hours later. At these times, in patients with a reduction of at least one point in VeXus, the furosemide infusion will be maintained. If there is a worsening or no improvement of at least one point in the VeXus, the infusion will be doubled.In patients where there are signs of hypoperfusion, furosemide therapy will be discontinued. The administration of furosemide will also be interrupted in patients who develop serum sodium > 160 mEq/L; metabolic alkalosis (bicarbonate > 35 mEq/L) or potassium < 3mEq/L. In patients randomized to the usual therapy group, the attending physician will decide whether to prescribe furosemide or not according to his assessment without any defined time criteria. All other aspects of care will be managed according to routine unit protocols

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Hospitalization in ICU for at least 48 hours.
* Patient in septic shock for at least 24 hours and clinically stable defined by mean arterial pressure ≥ 65 mmHg and maximum infusion of 0.20 μg/kg/min of norepinephrine and lactate < 4.0 mmol/L.
* Signed informed consent

Exclusion Criteria:

* Patients in use of more than one vasopressor
* Known right ventricle dysfunction
* Indication to use furosemide for other reasons
* Hypernatremia (Na >160 mmol/L)
* Advanced acute kidney injury(KDIGO 3)
* Current renal replacement therapy
* Anuria for ≥ 6 hours
* Hepatorenal syndrome
* Patients in palliative care
* Furosemide allergy.
* Rhabdomyolysis.
* Major burn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Hierarchy outcome: death in the ICU, need for renal replacement therapy during ICU stay and serum creatinine value on the third day after randomization | three days
  The outcome of the study will be assessed by the win rate ("Win ratio WR) between the intervention arm and the usual care arm defined by the occurrence in hierarchical order of one of the following events:
  * Death in ICU
  * Need for renal replacement therapy during ICU stay
  * Serum creatinine value on the third day after randomization

SECONDARY OUTCOMES:
fluid balance | three days
  fluid balance during the first three days
PaO2/FiO2 | three days
  worst PaO2/FiO2 during the first three days

OTHER OUTCOMES:
intervention stopping criteria: hypokalemia, hypernatremia and metabolic acidosis | Three days
  As safety outcomes, we will assess the following events potentially attributed to intervention: Na >160 mEq/L; metabolic alkalosis (bicarbonate> 35 mEq/L), potassium <3mEq/L

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Machado, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be provided upon request and after analysis of the study executive committee
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after 6 months of publication and for 5 years
Access Criteria: EC approval